CLINICAL TRIAL: NCT04856787
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II/III Study of SHR-1701 or Placebo in Combination With BP102 (Biosimilar to Bevacizumab) and XELOX in First-line Treatment of mCRC
Brief Title: A Clinical Studyf of SHR-1701 or Placebo in Combination With BP102 and XELOX in the First-line Treatment of mCRC
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Adjustment of the Company's R&D Strategy
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1701-III-301
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-1701 in combination with BP102 and XELOX（Phase 2） (Experimental)
  Interventions: Drug: SHR-1701、 BP102 、XELOX
- SHR-1701 in combination with BP102 and XELOX （Phase 3） (Experimental)
  Interventions: Drug: SHR-1701、 BP102 、XELOX
- placebo in combination with BP102 and XELOX (Placebo Comparator)
  Interventions: Drug: placebo、 BP102、 XELOX

INTERVENTIONS:
Drug: SHR-1701、 BP102 、XELOX — Phase 2：Single Group
  Drug:SHR-1701 30mg/kg，IV ,every 3 week
  Drug：BP102 7.5mg/kg，IV,every 3 week
  Drug: Oxaliplatin 130mg/m2 ，IV,every 3 week
  Drug:Capecitabine The total daily dose was 2000mg/m2, OR，Each cycle was administered for 2 consecutive weeks, followed by a week of rest, with a treatment cycle every 21 days
  Arms: SHR-1701 in combination with BP102 and XELOX（Phase 2）
Drug: SHR-1701、 BP102 、XELOX — Phase 3：Randomized
  Drug:SHR-1701 30mg/kg，IV ,every 3 week
  Drug：BP102 7.5mg/kg，IV,every 3 week
  Drug: Oxaliplatin 130mg/m2 ，IV,every 3 week
  Drug:Capecitabine The total daily dose was 2000mg/m2, OR，Each cycle was administered for 2 consecutive weeks, followed by a week of rest, with a treatment cycle every 21 days
  Arms: SHR-1701 in combination with BP102 and XELOX （Phase 3）
Drug: placebo、 BP102、 XELOX — Phase 3：Randomized
  Drug:Placebo 30mg/kg，IV ,every 3 week
  Drug：BP102 7.5mg/kg，IV,every 3 week
  Drug: Oxaliplatin 130mg/m2 ，IV,every 3 week
  Drug:Capecitabine The total daily dose was 2000mg/m2, OR，Each cycle was administered for 2 consecutive weeks, followed by a week of rest, with a treatment cycle every 21 days
  Arms: placebo in combination with BP102 and XELOX

SUMMARY:
This is a two-arm, randomized, double-blinded, multicenter phase II/III clinical study to evaluate the safety and clinical efficacy of SHR-1701 or placebo in combination with BP102 (biosimilar to bevacizumab) and XELOX in first-line treatment of patients with mCRC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable recurrent or metastatic adenocarcinoma of the colon or rectum confirmed histologically
2. For subjects who have not previously received any systemic antitumor therapy and who have previously received neoadjuvant or adjuvant therapy, the first detection of recurrence or metastasis should be ≥12 months after the last administration of neoadjuvant or adjuvant therapy
3. At least 1 measurable lesion according to RECIST V1.1
4. The vital organs are functioning well
5. ECOG score is 0 ~ 1
6. Contraception was initiated from the signing of the informed consent until at least 6 months after the last dosing of the study drug

Exclusion Criteria:

1. Recurrent or metastatic lesions can be treated with radical surgery
2. Presence of central nervous system or meningeal metastases;
3. Moderate and severe ascites of clinical symptoms;Uncontrolled or moderate or greater pleural effusion or pericardial effusion
4. Poorly controlled hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg in the case of regular antihypertensive therapy) and prior hypertensive crisis or hypertensive encephalopathy
5. Severe cardiovascular and cerebrovascular diseases;Have clinical heart symptoms or diseases that are not well controlledSubjects with a history of myocardial infarction or unstable angina pectoris
6. Subject with current interstitial pneumonia or interstitial lung disease, or with a previous history of interstitial pneumonia or interstitial lung disease requiring hormone therapy
7. Previous treatment with targeted T cell costimulatory molecules and immune checkpoint inhibitors;Previous treatment with antiepidermal growth factor receptor or any antiangiogenic drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Phase 2:ORR | up to 2 years
  Objective response rate (assessed by the investigators based on RECIST v1.1)
Phase 2:Incidence of Adverse Events (AEs) by CTCAE v5.0 | up to 2 years
  Assess safety and tolerability of SHR-1701 in combination with BP102 and XELOX
Phase 3:PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 2 years
  Progression-free survival (assessed by independent radiological review committee (IRRC) based on RECIST v1.1)

SECONDARY OUTCOMES:
DCR | up to 2 years
  Disease control rate，the proportion of patients with the best overall response of CR, PR, or stable disease (SD) 。
OS | up to 2 years
  Overall survival ，from the date of first dose unitl the date of death from any cause。
PFS | up to 2 years
  Progression-free survival from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed (assessed by independent radiological review committee (IRRC) based on iRECIST，by the investigators based on RECIST v1.1))。
Duration of response | up to 2 years
  Duration of response，from the date when CR or PR (whichever recorded earlier) is firstly achieved until the date when disease progression or death is firstly recorded (whichever occurs earlier),assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Qiu MZ, Bai Y, Wang J, Gu K, Yang M, He Y, Yi C, Jin Y, Liu B, Wang F, Chen YK, Dai W, Jiang Y, Huang C, Xu RH, Luo HY. Addition of SHR-1701 to first-line capecitabine and oxaliplatin (XELOX) plus bevacizumab for unresectable metastatic colorectal cancer. Signal Transduct Target Ther. 2024 Dec 16;9(1):349. doi: 10.1038/s41392-024-02063-0. PMID 39676137